CLINICAL TRIAL: NCT04015713
Title: LILAC - TB : Lowering InterLeukin-1 Receptor Antagonist Concentrations After TB Treatment Onset : a Proof of Concept Study in Cambodia and Ivory Coast (ANRS 12394)
Brief Title: Lowering InterLeukin-1 Receptor Antagonist Concentrations After TB Treatment Onset
Acronym: LILAC-TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut Pasteur, Cambodia (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS 12394 LILAC-TB
Record Dates: First submitted 2019-07-02; First posted 2019-07-11 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples drawn at inclusion, week 1, week 2, week 4 and week 8 and biobank (DBS, plasma and dry blood pellet)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TB HIV-negative: Patients will receive standard TB treatment and will be followed according to the national procedures.
  In addition, plasma samples will be collected at baseline, Week 1, Week 2, Week 4 and Week 8 to measure IL-1Ra, sCD163 and IP-10. Baseline will be the initiation of TB treatment.
  All participants will be followed 24 weeks.
- TB HIV-positive: Patients will receive standard TB treatment and will be followed according to the national procedures.
  In addition, plasma samples will be collected at baseline, Week 1, Week 2, Week 4 and Week 8 to measure IL-1Ra, sCD163 and IP-10. Baseline will be the initiation of TB treatment.
  All participants will be followed 24 weeks.

SUMMARY:
Despite marked improvements in the diagnosis of tuberculosis there are difficulties in diagnosing and monitoring treatment outcome among TB patients. The use of immunological biomarkers alone or in combination with other clinical parameters could predict early the response to TB treatment. The aim of this study is to demonstrate that the IL-1 receptor antagonist (IL-1Ra) concentrations significantly decrease within two weeks following TB treatment initiation in adults with active documented TB.

DETAILED DESCRIPTION:
The HIV/AIDS epidemic and Tuberculosis (TB) remain important challenges for global public health and are strongly linked. Despite marked improvements in the diagnosis of tuberculosis, there are difficulties in diagnosing and monitoring treatment outcome among TB patients. The use of immunological biomarkers alone or in combination with other clinical parameters could better predict the response to TB treatment. The aim of this study is to demonstrate that the IL-1 receptor antagonist (IL-1Ra) concentrations significantly decrease within two weeks following TB treatment initiation in adults with active documented TB. This is a proof-of-concept study, among 100 patients (50 HIV positive and 50 HIV negative) with documented active TB, in Cambodge and Côte d'Ivoire. Patients recruited for this study will receive the standard TB treatment per their respective national treatment guidelines. Plasma samples will be collected at baseline (initiation of TB treatment), weeks 1, 2, 4 and 8 to measure IL-1Ra, sCD163 and IP-10.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Evidence of TB, with: positive Xpert MTB/RIF
* For HIV infected patients:

  * ART-naïve
  * Regardless of CD4 cell counts
* Written informed consent
* Willingness to be followed up in the study clinics for 6 months after inclusion

Exclusion Criteria:

* Mycobacterium tuberculosis strain resistant to rifampin with Xpert MTB/RIF
* Ongoing TB treatment
* Overt evidence of other ongoing opportunistic infections
* Pregnant or breastfeeding women
* Karnofsky score ≤ 30
* Person unable to understand the study
* Person currently participating in clinical trial
* Females on oestroprogestative and progestative hormonal contraception

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 100 patients with documented active TB, 50 in Cambodia and 50 in Côte d'Ivoire
  * 60 patients HIV-infected and 40 patients HIV negative
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Evolution of the plasma concentration of IL-1Ra between baseline (initiation of TB treatment) and Week 2 | 2 weeks
  To measure plasma concentrations of IL - 1Ra among TB patients after two weeks of TB treatment

SECONDARY OUTCOMES:
Evolution of the plasma concentration of IL-1Ra between baseline (initation of TB treatment) and weeks 1, 2, 4 and 8 | 8 weeks
  To measure plasma concentrations of IL - 1Ra and assess the evolution of the concentration of IL-1Ra among TB patients at week 1, week 2, week 4 and week 8 after treatment initiation
Evolution of the concentration of sCD163 between baseline (initiation of TB treatment) and weeks 1, 2, 4 and 8 | 8 weeks
  To measure plasma concentrations of sCD163 and assess the evolution of the concentration of IL-1Ra among TB patients at week 1, week 2, week 4 and week 8 after treatment initiation
Evolution of the plasma concentration of IP-10 between baseline (initiation of TB treatment) and weeks 1, 2, 4 and 8 | 8 weeks
  To measure plasma concentrations of IP-10 and assess the evolution of the concentration of IL-1Ra among TB patients at week 1, week 2, week 4 and week 8 after treatment initiation
Impact of the occurrence of events on the evolution of biomarkers from baseline (initiation of TB treatment) to the end of treatment (Week 24) | 24 weeks
  Impact of the occurrence of the following events/situations on the evolution of biomarkers (IL-1Ra,sCD163 and IP-10) : intercurrent infection, TB-associated immune reconstitution inflammatory syndrome (IRIS), TB treatment outcome, MTb strains resistant to TB drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Weiss, MD,PhD, Principal Investigator — APHP Georges Pompidou European Hospital
Locations (2):
- Institut Pasteur Cambodge, Phnom Penh, Cambodia
- CEPREF/Programme PACCI, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No